CLINICAL TRIAL: NCT03184896
Title: Multicenter Prospective Observational Study in Hip Fracture Among Older Adults
Brief Title: Services Mapping Among Older Adults With Hip Fracture
Acronym: HiFit
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: The George Institute for Global Health, China (Other)
Collaborators: Beijing Hospital (Other Government); Beijing Anzhen Hospital (Other); Beijing Friendship Hospital (Other); Beijing Shuyi Hospital (Other); Beijing Fangshan District Liangxiang Hospital (Other); Beijing Changping District Hospital (Unknown); Beijing Jishuitan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 0281001
Record Dates: First submitted 2017-06-08; First posted 2017-06-14 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hip Fracture
  Interventions: Procedure: Hip Fracture Surgery

INTERVENTIONS:
Procedure: Hip Fracture Surgery — Hip Fracture Surgery

SUMMARY:
Hip fracture is a osteoporosis-related fracture with higher mortality, and is a major public health issue in China. The British Orthopedic Association and the British Geriatric Society have published the UK Blue Book, which summarizes current evidence and best practice in the hip fracture care and secondary prevention, but this kind of standardized practice in hip fracture care is not yet existed in China. The Blue Book standards will be used as the most contemporary evidence-based guidelines for management of hip fracture.This study is to prospectively examine the barriers and facilitators in the current management of hospital in China by comparing the Blue Book standards.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 65 years old or over;
* Hip fracture with X-ray-confirmed femoral neck, trochanteric or sub-trochanteric fracture;
* Within 21 days of a hip fracture;
* Willingness to sign informed consent form;

Exclusion Criteria:

* Patients with pathological fractures;
* With terminal malignancies.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients who have a history of an acute injury that occurred within 21 days, and diagosed by X-ray will be recruited in this study.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2018-11-14 (Actual); Primary Completion 2021-11-13 (Estimated); Study Completion 2021-11-13 (Estimated)

PRIMARY OUTCOMES:
Operative administration within 48 hours | One year
  The proportion of patients who are operated within 48 hours in the past one year

SECONDARY OUTCOMES:
A&E Admission within 4 hours | One year
  The proportion of patients who admit to orthopaedic ward from A&E within 4 hours in the past one year
The Incidence of Pressure Ulcer | One year
  The incidence of pressure ulcer in the past one year via nurses provide assessment
The Proportion of Patients Who Receive Geriatrician Assessment | One year
  The proportion of patients who receive the assessment of geriatricians in the past one year
The Proportion of Patients Who Receive Osteoporosis Assessment and Treatment | One year
  The proportion of patients who receive osteoporosis assessment and treatment the hospital provided in the past one year
The Proportion of Patients Who Receive Specialist Falls Assessment | One year
  The proportion of patients who receive specialist falls assessment in the past one year

OTHER OUTCOMES:
Mortality Rate in One Month, Four-Month, and One Year | One month, four-month, and one year
  The mortality rate in one, four-month, and one year after admission to hospital
The Incidence of Complications in One Month, Four-Month, and One year | One month, four-month, and one year
  The incidence of complications in one month, four-month and one year after admission to hospital, including pneumonia, deep vein thrombosis, heart disease, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- The George Institute, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu T, Zhang X, Zhang J, Ye P, Yang M, Tian M. Effect of the orthogeriatric co-management on older hip fracture patients with multimorbidity: a post-hoc exploratory subgroup analysis of a non-randomised controlled trial. J Orthop Surg Res. 2024 Nov 21;19(1):780. doi: 10.1186/s13018-024-05263-0. PMID 39574198